CLINICAL TRIAL: NCT02703545
Title: International CAPS Registry: Operated Cases and Cases With Advanced Disease Among High-risk Individuals Participating in a Pancreatic Cancer Surveillance Program; a Case-control Study
Brief Title: International CAPS Registry: Pancreas Cancer Cases in Surveillance Programs
Acronym: CAPS Registry
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00027287
Record Dates: First submitted 2015-07-16; First posted 2016-03-09 (Estimated); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Pancreas Cancer
Keywords: familial pancreas cancer; pancreatic cyst
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatic Cyst

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Peutz-Jeghers syndrome
- Familial pancreas cancer: at least 2 close relatives affected with pancreas cancer on same side of family
  1. first degree relative and 1 second degree relative(1st degree link) or
  2. first degree relatives or
  1 first degree relative and 2 or more second degree relatives
- Germline mutation Carrier 10 % risk: BRCA2 mutation carrier with family history of pancreas cancer or, PALB2 mutation carrier or, FAMMM (p16/CDKN2A) mutation carrier
- Germline mutation carrier 5 % risk: BRCA1 mutation carrier with family history of pancreas cancer or, HNPCC (Lynch Syndrome) with family history of pancreas cancer or, ATM gene mutation
- Hereditary pancreatitis: PRSS1, PRSS2, CTRC gene mutations

SUMMARY:
Various centers around the world are currently investigating the feasibility and yield of surveillance for pancreatic cancer in high-risk individuals. Evidence is beginning to accumulate that surveillance may lead to the early detection of non-invasive precursor lesions and asymptomatic early stage cancer. Ultimately, the goal of surveillance is to reduce mortality in these high risk individuals, but before this can be confirmed many research questions need to be answered. While the numbers of high-risk individuals screened in each separate screening facility are likely too small to properly address many of these questions, pooling data comprises a sizable sample size providing unique research opportunities. The objective of this study is retrospectively review all cases of high-risk individuals participating in our pancreatic surveillance program in whom 1) a suspicious precursor lesions was detected for which a pancreatic resection was performed and 2) in whom an advanced malignant disease was diagnosed. The de-identified information will be entered into an international multicenter database registry.

DETAILED DESCRIPTION:
The study is a retrospective review of all cases of high-risk individuals participating in our pancreatic surveillance program in whom 1) a suspicious precursor lesions was detected for which a pancreatic resection was performed and 2) in whom an advanced malignant disease was diagnosed. The de-identified information will be entered into an international multicenter database registry.

ELIGIBILITY:
Inclusion Criteria:

* Elevated pancreas cancer risk cohort with pancreas cancer or dysplastic pancreas changes

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Familial or genetic pancreas cancer risk cohorts found to have pancreas cancer or pancreas dysplasia
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Proportion of patients and resected lesions with pancreatic cancer in situ (high grade dysplasia) or invasive malignancy | 5 years
  Prevalence of pancreatic neoplasia high risk patients who had surgery for detected lesions in screening programs

SECONDARY OUTCOMES:
Indications for pancreas surgery | 5 years
  Pathology or imagining related to surgery indication
Proportion of specific types of pancreatic neoplasms by lesion type | 5 years
Incidence of pancreatic in-situ and invasive malignancy after baseline screening | 5 years
  Proportion of patients who had surgery or biopsy for new pancreatic lesions on follow-up
Calculate all-cause and disease specific mortality | 5 years
Calculate survival time from point of diagnosis and treatment | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Marcia I Canto, MD, Principal Investigator — Johns Hopkins University

REFERENCES:
- [Result] Canto MI, Harinck F, Hruban RH, Offerhaus GJ, Poley JW, Kamel I, Nio Y, Schulick RS, Bassi C, Kluijt I, Levy MJ, Chak A, Fockens P, Goggins M, Bruno M; International Cancer of Pancreas Screening (CAPS) Consortium. International Cancer of the Pancreas Screening (CAPS) Consortium summit on the management of patients with increased risk for familial pancreatic cancer. Gut. 2013 Mar;62(3):339-47. doi: 10.1136/gutjnl-2012-303108. Epub 2012 Nov 7. PMID 23135763
- [Result] Goggins M, Overbeek KA, Brand R, Syngal S, Del Chiaro M, Bartsch DK, Bassi C, Carrato A, Farrell J, Fishman EK, Fockens P, Gress TM, van Hooft JE, Hruban RH, Kastrinos F, Klein A, Lennon AM, Lucas A, Park W, Rustgi A, Simeone D, Stoffel E, Vasen HFA, Cahen DL, Canto MI, Bruno M; International Cancer of the Pancreas Screening (CAPS) consortium. Management of patients with increased risk for familial pancreatic cancer: updated recommendations from the International Cancer of the Pancreas Screening (CAPS) Consortium. Gut. 2020 Jan;69(1):7-17. doi: 10.1136/gutjnl-2019-319352. Epub 2019 Oct 31. PMID 31672839